CLINICAL TRIAL: NCT06476288
Title: Feasibility and Acceptability of Remote Ischemic Conditioning to Achieve High-Intensity Rehabilitation Effects and Increase Resilience in Older Individuals
Brief Title: RIC (Remote Ischemic Conditioning) in Older Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00115014
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Old Age; Mobility Limitation; Debility
Keywords: Exercise; Strength training; Conditioning; RIC; Remote Ischemic Conditioning; Ischemic Conditioning
MeSH Terms: conditions — Mobility Limitation; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be split into two different groups: one receiving a high-dose RIC intervention with low-intensity exercise and the other receiving a low-dose RIC intervention with low-intensity exercise. The assignment to the two different groups will be done by a computer in a process similar to flipping a coin in a 1:1 ratio. There will be 10 participants in each group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose RIC (Remote Ischemic Conditioning) Intervention (Active Comparator): Low-intensity resistance exercise training plus high-dose RIC.
  Interventions: Other: Low-intensity resistance exercise training; Other: High-Dose Remote ischemic conditioning (RIC)
- Low-Dose RIC Intervention (Placebo Comparator): Low-intensity resistance exercise training plus low-dose RIC.
  Interventions: Other: Low-intensity resistance exercise training; Other: Low-Dose Remote ischemic conditioning (RIC)

INTERVENTIONS:
Other: Low-intensity resistance exercise training — The intervention protocol will consist of 60 minutes of low-intensity resistance exercise training 3x/week for 6 weeks.
Other: High-Dose Remote ischemic conditioning (RIC) — Treatment dose of RIC- the RIC cuff will be inflated to 20 mmHg over the participant's systolic blood pressure. The treatment dose of RIC will be applied in 4 sets of cycles with inflating the cuff and leaving it pumped for 5 minutes then deflating the cuff for an off period of 5 minutes. Total treatment time will be 35 minutes.
  Arms: High-Dose RIC (Remote Ischemic Conditioning) Intervention
Other: Low-Dose Remote ischemic conditioning (RIC) — This dose will be the control for the study. Low-dose RIC- the RIC cuff will be inflated to 10 mmHg below the participant's diastolic blood pressure. The low-dose RIC will be applied in 4 sets of cycles with inflating the cuff and leaving it pumped for 5 minutes then deflating the cuff for an off period of 5 minutes. Total treatment time will be 35 minutes.
  Arms: Low-Dose RIC Intervention

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a technique called remote ischemic conditioning (RIC) that aims to improve muscle strength, muscle mass, exercise tolerance, resilience (i.e. how well someone responds to a stressor), quality of life, physical activity, and physical function when added to rehabilitative exercise training in individuals over age 65 who have some difficulty with mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 65 years and referred to an exercise program for functional decline, deconditioning, or fall risk
2. Exercises ≤ 2x/week on a regular interval

Exclusion Criteria:

1. Unstable heart disease as determined by the investigator or study physician
2. History of any orthopaedic, neurologic, or metabolic condition that would contraindicate exercise testing/training as determined by the investigator
3. Cognitive inability to follow directions and safely participate in exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study intervention as measured by the number of participants who completed the study | Up to 6 weeks
Feasibility of study intervention as measured by the attrition rate | Up to 6 weeks
  Attrition rate is expressed as a percentage and is calculated by dividing the number of non-completers by the total number of participants.
Feasibility of study intervention as measured by the number of exercise visits attended per participant | Up to 6 weeks
Feasibility of study intervention as measured by the number of RIC home applications completed per participant | Up to 6 weeks
Acceptability of study intervention as measured by an Intervention Acceptability Questionnaire | Up to 6 weeks
  Each participant will complete an Intervention Acceptability Questionnaire with responses on a 5-point Likert scale, where a higher score indicates greater acceptability.

SECONDARY OUTCOMES:
Feasibility of collecting blood samples during study as measured by the success rate of collection | Up to 6 weeks
Change in Short Physical Performance Battery (SPPB) | Baseline to post-intervention visit (approximately 7 weeks)
  The SPPB measures changes in physical function.
Change in muscle strength as measured by dynamometry | Baseline to post-intervention visit (approximately 7 weeks)
  Measurements made with isokinetic dynamometry, hand-held dynamometry and DXA scans completed at pre- and post-intervention.
Change in exercise tolerance as measured by VO2peak testing | Baseline to post-intervention visit (approximately 7 weeks)
Change in quality of life as measured by PROMIS-29 | Baseline to post-intervention visit (approximately 7 weeks)
Change in Brief Resilience 5-point Likert Scale | Baseline to post-intervention visit (approximately 7 weeks)
  Higher score indicates greater resilience.
Change in vascular function as measured by arterial tonometry | Baseline to post-intervention visit (approximately 7 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: W Todd Cade, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No